CLINICAL TRIAL: NCT01068561
Title: Phase 1 Study Of Autologous Bone Marrow-Derived Stem Cells Transplantation For Retinitis Pigmentosa
Brief Title: Autologous Bone Marrow-Derived Stem Cells Transplantation For Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rubens Camargo Siqueira, MD,PhD, University of Sao Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPRS
Record Dates: First submitted 2010-02-10; First posted 2010-02-15 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; stem cell; bone marrow
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test group (Experimental): open-label study of retinitis pigmentosa patients with best-corrected visual acuity (BCVA) worse than 20/200.
  Interventions: Biological: intravitreal injection of autologous bone marrow stem cells

INTERVENTIONS:
Biological: intravitreal injection of autologous bone marrow stem cells — One intravitreal injection of a 0.1-ml cell suspension containing around 10x106 bone marrow mononuclear stem cells(BMMSC). All treatments were performed by a single retinal specialist using topical proparacaine drops under sterile conditions (eyelid speculum and povidone-iodine). Autologous BMMSC were injected into the vitreous cavity using a 27 gauge needle inserted through the inferotemporal pars plana 3.0 - 3.5 mm posterior to the limbus. After the injection, central retinal artery perfusion was confirmed with indirect ophthalmoscopy. Patients were instructed to instill one drop of 0.3% ciprofloxacin into the injected eye four times daily for 1 week after the procedure.
  Other Names: Autologous bone marrow mononuclear stem cells

SUMMARY:
The purpose of this study is to evaluate the short-term safety of a single intravitreal injection of autologous bone marrow stem cells in patients with retinitis pigmentosa.

DETAILED DESCRIPTION:
A prospective phase I, nonrandomized open-label study of retinitis pigmentosa patients with best-corrected ETDRS visual acuity (BCVA) worse than 20/200. Standardized ophthalmic evaluation will be perform at baseline and at weeks 1, 4,12 and 24 (±1) following intravitreal injection of 10 x 106 bone marrow stem cells/ 0,1ml . Three measures will be used to evaluate the short-term safety of intravitreal of ABMDSC: 1) severe visual loss, defined as a drop in 15 letters on ETDRS visual acuity scale; 2) decrease in ERG response; 3) decrease in 5 square degrees on visual field; secondary safety outcomes : 1) increase in intra-ocular inflammation defined herein as anterior chamber cells and flare higher than 3+ for more than 1 month after injection according to a classification described elsewhere ; 2) decrease in CMT more than 50um; 3)genesis of abnormal tissues (teratomas) or tumors; 4) qualitative changes in retinal or choroidal perfusion, like macular nonperfusion. Secondary outcome measures will be used to evaluate the short-term efficiency of intravitreal of ABMDSC: 1) improvement in ERG response; 2) increase in visual field: 3) increase in CSMT > 50um and not related to macular edema; 4) increase > 5 letters on BCVA

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of retinitis pigmentosa
* logarithm of minimum angle of resolution (logMAR) BCVA of 1.0 (Snellen equivalent, 20/200) or worse

Exclusion Criteria:

* previous ocular surgery other than cataract
* presence of cataract or other media opacity that would influence ocular fundus documentation and adequate ERG and visual field evaluation
* other ophthalmic disease like glaucoma and uveitis
* previous history of blood disorders like leukemia
* known allergy to fluorescein or indocyanine green
* known coagulation abnormalities or current use of anticoagulative medication other than aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
severe visual loss, defined as a drop in 15 letters on ETDRS visual acuity scale | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rubens C Siqueira, MD,PhD, Principal Investigator — Research Center Rubens Siqueira,Catanduva Medicine School and São Paulo University
Locations (1):
- CPRS, São Jose Do Rio Preto, São Paulo, Brazil